CLINICAL TRIAL: NCT00148499
Title: Efficacy and Tolerability of Ambroxol Lozenge 20 mg in Relieving Pain of Sore Throat in Patients With Acute Viral Pharyngitis-A Randomised, Double-blind,Placebo- and Active-controlled Parallel Group Study
Brief Title: Efficacy and Tolerability of Ambroxol Lozenge 20 mf in Relieving Pain of Sore Throat in Pat. With Acute/Viralpharyngitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18.489
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Benzocaine

INTERVENTIONS:
Drug: Ambroxol hydrochloride (Mucoangin?)
Drug: benzocaine

SUMMARY:
The purpose of this trial is to investigate efficacy and tolerability of lozenges containing 20 mg a mbroxol hydrochloride (Mucoangin?) relative to lozenges containing placebo and lozenges containing 3 mg benzocaine in relieving pain of sore throat in patients suffering from acute viral pharyngitis.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo- and active-controlled parallel group study in adult pat ients, suffering from acute viral pharyngitis and throat pain of at least moderate intensity.

The whole study will last for up to 4 days, on each of test days patients will take one lozenge cont aining Ambroxol hydrochlorid 20 mg/ or placebo/ or benzocaine lozenge 3 mg up to 6 lozenges per day.

Using Patient Diaries the assessment of tolerability and efficacy by the patient will be obtained.

Study Hypothesis:

The primary hypothesis to be tested is the test of superiority of ambroxol 20 mg in comparison to placebo. If and only if the corresponding test of superiority to placebo is statistically significant, the hypothesis of non-inferiority of am broxol 20 mg in comparison to benzocaine 3 mg will be tested.

Comparison(s):

For the primary comparison the placebo lozenges will be used, for the secondary comparison the benzocaine 3 mg lozenges will be used.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients having a sore throat with acute viral pharyngitis.
2. Female and male patients between the ages of 18 and 80 years.
3. The throat pain intensity is rated at least moderate on the VRS (PI).
4. Written Informed Consent is given by the patient.
5. Compliance by the patient seems guaranteed, and patient seems to be able to understand and complete the patient diary.
6. Patient able to remain at the doctor's practice for the initial 3 hours follo wing the first intake of study medication, and able to return for the study visi ts.

EXCLUSION CRITERIA

1. Female patients of child-bearing potential that are:

   1. Pregnant
   2. Currently breastfeeding
   3. NOT practicing acceptable methods of birth control, or NOT planning to contin ue practicing an acceptable method throughout the study. Acceptable methods of birth control include surgical sterilisation, intra uterine device, oral, implan table, injectable contraceptives or double-barrier method.
2. Patients with symptoms of primarily bacterial pharyngitis or bacterial secon dary infection (clinical findings inter alia assessment of exudate).
3. First indication of symptoms of acute pharyngitis (e.g. sore throat) occurre d more than 3 days ago.
4. Patients who suffered from acute viral or bacterial pharyngitis in the past 4 weeks.
5. Patient who in the past week, or during the study will require treatment with the following: antibiotics steroids for oral, inhaling or topical application expectorants or antitussives. No physical therapy (e.g. throat compress, throa t rinsing) may be applied during the trial. Patients who have used analgesics or anti-inflammatory agents less than two half-lives of the applicable drug before study entry, or who will require their use in the 3 hours after taking the firs t lozenge.
6. Patients with mouth breathing as a result of nasal congestion.
7. Known hypersensitivity to Ambroxol or to auxiliary substances contained in t he lozenge.
8. Existing tumour condition currently under treatment.
9. Alcohol, and/or drug abuse.
10. Any clinical condition which, in the opinion of the investigator would not a llow safe completion of the protocol and safe administration of trial medication.
11. Any investigational therapy within 30 days prior to randomisation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06

PRIMARY OUTCOMES:
Primary Endpoint: Time-weighted average of the pain intensity difference from pre-dose baseline over the first 3 hours after the first lozenge expressed as a ratio of the pre-dose baseline (SPIDnorm)

SECONDARY OUTCOMES:
Pain intensity (PI) and pain intensity difference from pre-dose baseline (PID) Time to onset of action after the first lozenge Assessment of efficacy Assessment of tolerability by the patient and investigator Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BI Pharma Ges mbH Wien
Locations (12):
- Romania (2):
  - Medicover, Bucharest
  - Victor Babes Clincial Hospital, Bucharest
- Ukraine (10):
  - Regional Student Hospital, Kharkiv
  - Regional Clinical Hospital, Kharkiv
  - City Clinical Otolaryngological Hospital, Kharkiv
  - City Clinical Hospital No. 17, Kharkiv
  - City Clinical Hospital No. 11, Kharkiv
  - City Clinical Hospital No. 26, Kharkiv
  - Academy of Medical Science named after O.S. Kolomyichenko, Kiev
  - City Clinical Hospital No. 9, Kiev
  - City Clinical Hospital No. 11, Odesa
  - Regional Clinical Hospital, Zaporizhzhya

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/19137906